CLINICAL TRIAL: NCT00810771
Title: Evaluating a Preference-based Intervention for Increasing CRC Screening
Brief Title: Evaluating a Preference-based Intervention for Increasing Colorectal Cancer Screening
Acronym: EPIIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 06-205
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Neoplasms
Keywords: Hospitals, Veterans; Mass Screening/utilization; Patient Preference; Prevention & Control; Epidemiology
MeSH Terms: conditions — Colorectal Neoplasms; Patient Acceptance of Health Care; Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Preference-tailored (PT) intervention (Experimental): Intervention:
  Behavioral: Standard Information Behavioral: Preference-tailored Information
  Interventions: Behavioral: Standard Information; Behavioral: Preference-tailored Information
- Standard information (SI) intervention (Active Comparator): Behavioral: Standard Information
  Interventions: Behavioral: Standard Information
- Usual Care (No Intervention): Due to budget and time constraints this group was not powered as a true study arm but was used to assess the impact of our baseline physician information letter and to control for any other interventions of system-wide initiatives that may occur during the study timeframe and impact rated of CRC screening. Data was not collected on every participant in this arm.

INTERVENTIONS:
Behavioral: Standard Information — A computer based educational overview of CRC and CRC test options will be presented to the subject. The subject will be given a handout with a brief description of each of the screening options and will include the test that they have chosen as their preferred test. The subjects will be asked to take this handout to their upcoming clinic appointment and to discuss the screening options with their care provider.
  Arms: Preference-tailored (PT) intervention; Standard information (SI) intervention
Behavioral: Preference-tailored Information — A preference elicitation exercise that will generate a list of the three top attributes for the subject and the CRC screening test most consistent with these attributes. Subjects will be provided with a handout to take to their clinic appointment as the Standard Information group does, but with the addition of a listing of their top attributes and the test most consistent with their top attributes.
  Arms: Preference-tailored (PT) intervention

SUMMARY:
The goal of this study is to evaluate whether an educational tool about colorectal cancer (CRC) completed on a computer that helps patients clarify their CRC screening preferences will lead to increased screening rates for CRC compared to standard information delivered via computer.

DETAILED DESCRIPTION:
Background: Colorectal cancer (CRC) is a significant and preventable disease, yet CRC screening remains one of the lowest quality indicators in the VA healthcare system. Moreover, a recent VA directive recommends that CRC screening among Veterans should be based on their preferences, given that there is insufficient evidence to support recommending one test. However the impact of such a preference-based strategy on important outcomes, including screening adherence and cost, is unknown.

Objectives: The broad hypothesis of the proposed study is that helping Veterans clarify their CRC screening preferences will lead to increased adherence. The framework conceptualizes that preference clarification leads to more informed decision-making and, eventually, to better adherence with screening. The specific aims are: 1) To test the effectiveness of a preference-tailored (PT) vs. standard information (SI) intervention for increasing Veterans' CRC screening adherence; 2) To assess the impact of the intervention on informed decision making, knowledge and attitudes toward screening, decisional outcomes, and intention to get screened; and 3) To conduct a cost effectiveness analysis of the PT intervention for increasing CRC screening across the VA.

Methods: A randomized controlled trial of the PT vs. SI decision tool will be conducted in the Ann Arbor and Pittsburgh VA healthcare systems. The intervention was developed by the PI working with the Center for Health Communication Research at the University of Michigan. Eligible patients will be 552 (276 per group) Veterans between 50 and 78 who are due for CRC screening, and who have a primary care visit scheduled within the upcoming 4-6 weeks. Those at high risk (e.g., family or personal history of CRC) will be excluded. Providers will be informed of the study via regular mail and email. In Ann Arbor providers will be given the opportunity to opt-out their participants if they choose to do so. In Pittsburgh providers will be given lists of their participants as they are being considered for the study and will be given the chance to remove any potential participants from the contact list. Potential participants will be mailed an introductory letter. Those who do not opt-out will contacted by telephone. Participants will come to their primary care visit 40 minutes early, at which time they will complete informed consent. The intervention will be delivered via the Internet, and participants will be randomized to the PT or SI arm at the time of log-in. Study measures are consistent with the conceptual framework and based on the Preventive Health Model. Preference information will be collected through the computer program. Secondary outcomes and independent variables will be collected via telephone survey 3 days following the intervention. Adherence to screening will be collected from medical charts at 6 months. CRC screening information in a sub-sample of 80 Ann Arbor Veterans, not in either the PT or SI groups, will also be collected to measure "usual care" (UC). Pittsburgh will use the External Peer Review Program (EPRP) for the collection of clinical performance measures, more specifically CRC screening rates, to serve as an effective substitute for the UC group. Hypotheses related to each aim will be tested using multi-level modeling to control for between-provider effects. The overall hypothesis is that patients in the PT group will have higher rates of adherence to CRC screening at the 6 month follow-up point. Cost effectiveness analysis will determine whether a preference-based screening strategy could be cost effective for the VA healthcare system. The PI will work with the investigative team to disseminate the results through local and national VA websites, publications and presentations.

Status: Active, not recruiting.

ELIGIBILITY:
Inclusion Criteria:

* Clinic appointment at Ann Arbor or Pittsburgh VA during recruitment period.
* Age 50-78.
* Not up to date with CRC screening according to VA and USPSTF guidelines.
* At average risk for CRC (no history of CRC, adenomatous colon polyps, inflammatory bowel disease, and no family history of CRC).
* Has current address and telephone number listed in medical record.

Exclusion Criteria:

* DNR/DNI code status.
* Metastatic cancer.
* Stage D congestive heart failure.
* Severe COPD.
* Coronary artery disease (CAD) and MI within one year or CAD and unstable angina within 6 months.
* Dementia.
* Inability to conduct activities of daily living.
* Life expectancy less than one year.
* Other - anything else that limits CRC screening options.
* Scheduled for a colonoscopy, sigmoidoscopy, DCBE, or CTC.
* prior participation in this study
* unable to contact after 2 introductory letters (at least 6 months apart)

Ages: 50 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah T Hawley, PhD MPH BA, Principal Investigator — Ann Arbor VA Medical Center
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Center for Health Equity Research and Promotion, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Usual Care group is not counted toward the Enrollment total. See description of group below for additional details.
Pre-assignment Details: The Usual Care group is not counted toward the Enrollment total. See description of group below for additional details.
Groups:
- Preference-tailored (PT) Intervention: Standard Information: A computer based educational overview of CRC and CRC test options was presented to the subject. The subject was given a handout with a brief description of each of the screening options and which included the test that they have chosen as their preferred test. The subjects were asked to take this handout to their upcoming clinic appointment and to discuss the screening options with their care provider.
  Preference-tailored Information: A preference elicitation exercise generated a list of the three top attributes for the subject and the CRC screening test most consistent with these attributes. Subjects were provided with a handout to take to their clinic appointment as were the Standard Information group, but with the addition of a listing of their top attributes and the test most consistent with their top attributes.
- Standard Information (SI) Intervention: Standard Information: A computer based educational overview of CRC and CRC test options was presented to the subject. The subject was given a handout with a brief description of each of the screening options and which included the test that they have chosen as their preferred test. The subjects were asked to take this handout to their upcoming clinic appointment and to discuss the screening options with their care provider.
- Usual Care: Due to budget and time constraints this group is not powered as a true study arm but is being used to assess the impact of our baseline physician information letter and to control for any other interventions of system-wide initiatives that may have occurred during the study timeframe and impact rated of CRC screening.
Period: Overall Study
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention | Usual Care
Started | 232 | 234 | 84
Completed | 232 | 234 | 84
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants in Arm 1 and 2 reflect the number completing the survey. Not all participants enrolled to these arms completed the survey. Arm 3, "usual care" arm, was not a true 3rd arm and participants in this group did not complete the survey.
Groups:
- Preference-tailored (PT) Intervention: Preference-tailored Information: A preference elicitation exercise generated a list of the three top attributes for the subject and the CRC screening test most consistent with these attributes. Subjects were provided with a handout to take to their clinic appointment as were the Standard Information group, but with the addition of a listing of their top attributes and the test most consistent with their top attributes.
- Total: Total of all reporting groups
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention | Usual Care | Total
Number analyzed (Participants) | 198 | 197 | 84 | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 155 | 147 | 68 | 370
  >=65 years | 43 | 50 | 16 | 109
Age, Continuous [Mean (Full Range); unit: Years] | 60.1 [50 to 79] | 60.6 [50 to 79] | 59.5 [50 to 78] | 60.35 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 3 | 18
  Male | 194 | 186 | 81 | 461
Region of Enrollment [Number; unit: participants]
  United States | 198 | 197 | 84 | 479

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer (CRC) Screening Rate.
Description: The CRC Screening rate reports percentage of participant adherence with any Colorectal Cancer Screening test within 6 months of Decider Guider intervention. Decider Guider is a tool to help patients make an informed choice about colon cancer testing.
Time Frame: Within 6 months of Decider Guider intervention.
Measure: Number; unit: percentage of participants
Groups:
- Preference-tailored (PT) Intervention: Preference-tailored (PT) intervention
  Intervention:
  Behavioral: Standard Information Behavioral: Preference-tailored Information
  Preference-tailored Information: A preference elicitation exercise that will generate a list of the three top attributes for the subject and the CRC screening test most consistent with these attributes. Subjects will be provided with a handout to take to their clinic appointment as the Standard Information group does, but with the addition of a listing of their top attributes and the test most consistent with their top attributes.
- Standard Information (SI) Intervention: Standard information (SI) intervention
  Behavioral: Standard Information
  Standard Information: A computer based educational overview of CRC and CRC test options will be presented to the subject. The subject will be given a handout with a brief description of each of the screening options and will include the test that they have chosen as their preferred test. The subjects will be asked to take this handout to their upcoming clinic appointment and to discuss the screening options with their care provider.
- Usual Care: "Usual Care" - due to budget and time constraints this group is not powered as a true study arm but is being used to assess the impact of our baseline physician information letter and to control for any other interventions of system-wide initiatives that may have occurred during the study timeframe and impact rated of CRC screening.
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention | Usual Care
Number analyzed (Participants) | 232 | 234 | 84
percentage of participants | 40.1 | 40.2 | 19.3

2. Secondary Outcome: Number of Elements of Braddock's Informed Decision Making (IDM) Model Discussed With Provider
Description: Outcome measure using 6 items measuring degree of participation in IDM. Scaled and recategorized into Low, Moderate and High level of IDM. The range is from 1 (low level of IDM) to 6 (high level of IDM).
Time Frame: 3-5 days after Decider Guider intervention
Population: Data was not collected for Usual Care arm.
Measure: Mean (Full Range); unit: Degree of participation
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention
Number analyzed (Participants) | 198 | 197
Degree of participation | 5.72 [1 to 6] | 5.70 [1 to 6]
Statistical Analysis 1: Comparison: Preference-tailored (PT) Intervention vs Standard Information (SI) Intervention; Test type: Superiority or Other; p = 0.873, Chi-squared

3. Secondary Outcome: Colorectal Cancer Screening (CRCS) Knowledge and Attitudes.
Description: Outcome measure measuring knowledge of CRCS using 8-item knowledge measure (all true/false questions) developed for study, scaled and categorized into low/moderate/high knowledge, where low = low knowledge and high = high knowledge.
Time Frame: 3-5 days after Decider Guider intervention.
Population: Data was not collected for Usual Care arm.
Measure: Number; unit: percentage of participants
Groups:
- Preference-tailored (PT) Intervention: Preference-tailored (PT) intervention
  Intervention:
  Behavioral: Standard Information Behavioral: Preference-tailored Information
- Standard Information (SI) Intervention: Standard information (SI) intervention
  Behavioral: Standard Information
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention
Number analyzed (Participants) | 198 | 197
percentage of participants
  Low | 13.1 | 14.9
  Moderate | 66.2 | 67.7
  High | 20.7 | 17.4
Statistical Analysis 1: Comparison: Preference-tailored (PT) Intervention vs Standard Information (SI) Intervention; Test type: Superiority or Other; p = 0.671, Chi-squared

4. Secondary Outcome: Decisional Satisfaction
Description: Outcome measures measuring decisional satisfaction using 7-item scale categorized into low, moderate, high.
  Decisional satisfaction is a measure that was first developed by Margaret Holmes Rover and colleagues (Med Decis Making. 1996 Jan-Mar;16(1):58-64) to assess the perspective of a patient involved in a medical decision with the decision making process. The measure includes questions related to overall satisfaction, and satisfaction with the amount of information received, involvement in, degree of consistency with values, and time to make the decision. The measure includes 5 questions each on a 5 point scale where higher scores = higher satisfaction. When scaled into one overall measure of decision satisfaction, lower scores = lower satisfaction and higher scores = higher satisfaction.
Time Frame: 3-5 days after Decider Guider intervention.
Population: Data was not collected for Usual Care arm.
Measure: Number; unit: Percentage of participants
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention
Number analyzed (Participants) | 198 | 197
Percentage of participants
  Low | 16.6 | 29.4
  Moderate | 35.4 | 22.8
  High | 48 | 47.7
Statistical Analysis 1: Comparison: Preference-tailored (PT) Intervention vs Standard Information (SI) Intervention; Test type: Superiority or Other; p = 0.002, Chi-squared

5. Secondary Outcome: Intent to Get Colorectal Cancer Screening.
Description: Outcome measure measuring intent to get CRC screening using 5-item stage of readiness scale. Intent is measured by looking at the highest 2 items (I think I will get screened and I am committed to getting screened).
Time Frame: 3-5 days after Decider Guider intervention.
Population: Data was not collected for Usual Care arm.
Measure: Number; unit: percentage of participants
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention
Number analyzed (Participants) | 198 | 197
percentage of participants | 76.8 | 72.6
Statistical Analysis 1: Comparison: Preference-tailored (PT) Intervention vs Standard Information (SI) Intervention; Test type: Superiority or Other; p = 0.186, Chi-squared

6. Secondary Outcome: Self Efficacy.
Description: Outcome measure measuring self-efficacy using 5-item measure, dichotomized into low vs. high self-efficacy (confidence) in getting screened.
Time Frame: 3-5 days after Decider Guider intervention.
Population: Data was not collected for Usual Care arm.
Measure: Number; unit: percentage of participants
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention
Number analyzed (Participants) | 198 | 197
percentage of participants
  Low | 64.1 | 61.4
  High | 35.9 | 38.6
Statistical Analysis 1: Comparison: Preference-tailored (PT) Intervention vs Standard Information (SI) Intervention; Test type: Superiority or Other; p = 0.576, Chi-squared

7. Secondary Outcome: If Colorectal Cancer Screening Screening (CRCS) Discussed With Provider.
Description: Outcome measure measuring percentage of participants discussing CRCS with provider using single question (yes/no): "did you discuss Colorectal Cancer Screening with your provider?"
Time Frame: 3-5 days after Decider Guider intervention.
Population: Data was not collected for Usual Care arm.
Measure: Number; unit: percentage of participants
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention
Number analyzed (Participants) | 198 | 197
percentage of participants | 65.1 | 67.4
Statistical Analysis 1: Comparison: Preference-tailored (PT) Intervention vs Standard Information (SI) Intervention; Test type: Superiority or Other; p = 0.35, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Description: All Serious Adverse Events were determined by the IRB to be unrelated to study participation.
Groups:
- Preference-tailored (PT) Intervention: Preference-tailored (PT) intervention
- Standard Information (SI) Intervention: Standard information (SI) intervention
- Usual Care: "Usual Care" - due to budget and time constraints this group was not powered as a true study arm but was used to assess the impact of our baseline physician information letter and to control for any other interventions of system-wide initiatives that may occur during the study timeframe and impact rated of CRC screening. Data was not collected on every participant in this arm.
Arm/Group | Preference-tailored (PT) Intervention | Standard Information (SI) Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 3/232 | 3/234 | 0/84
Other Adverse Events (participants affected / at risk) | 0/232 | 0/234 | 0/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preference-tailored (PT) Intervention (N=232) | Standard Information (SI) Intervention (N=234) | Usual Care (N=84)
Hospitalization for Deep Venous Thrombus (DVT) and Abdominal Aortic Aneurysm (AAA) (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — The IRB determined this SAE to be unrelated to study participation.
Hospitalization for Acute Renal Failure and Diastolic Heart Failure. (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — The IRB determined this SAE to be unrelated to study participation.
Emergency room visit for atrial flutter; death 53 days later noted in chart, cause unknown (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — The IRB determined this SAE to be unrelated to study participation.
Hospitalization for esophageal cancer. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — The IRB determined this SAE to be unrelated to study participation.
Hospitalization for depression and alcohol intoxication (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — The IRB determined this SAE to be unrelated to study participation.
Death due to myocardial infarction. (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — The IRB determined this SAE to be unrelated to study participation.

LIMITATIONS AND CAVEATS:
Usual care arm was not true 3rd arm. We identified pts meeting eligibility criteria & randomized ~ 10th pt to be followed, measuring CRC screening 6 mos later. No intervention or survey. Only 79.6% of those enrolled completed survey.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes